CLINICAL TRIAL: NCT02862938
Title: A Randomized, Sham Controlled, Masked Phase II Study to Evaluate the Safety and Efficacy of Intravitreal Implantation of NT-501 Encapsulated Cell Therapy for the Treatment of Glaucoma
Brief Title: Study of NT-501 Encapsulated Cell Therapy for Glaucoma Neuroprotection and Vision Restoration
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Jeffrey L Goldberg, Professor and Chair of Ophthalmology, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 37202
Record Dates: First submitted 2016-08-01; First posted 2016-08-11 (Estimated); Last update posted 2025-11-04 (Actual); Status verified 2025-11

CONDITIONS: Glaucoma
MeSH Terms: conditions — Glaucoma | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NT-501 ECT Implant (Experimental): On eligible participants that are randomized to this group, the NT-501 Investigational product will be implanted in the study eye, and participants will be followed for 24 months.
  The investigational treatment, NT-501 ECT, provides intravitreal sustained release of soluble ciliary neurotrophic factor (CNTF) receptor after intraocular implantation.
  Interventions: Drug: NT-501 ECT implant
- Sham (Sham Comparator): To maintain masking, participants randomized to this group receive sham surgery and will be followed for 12 months. Following analysis of the 6 month data, if the open label extension (OLE) is not triggered, patients in the control group will continue on the original study schedule timeline trough month 24. If OLE is triggered participants will be offered the NT-501 ECT investigational product and will followed for additional 12 months.
  Interventions: Other: Sham

INTERVENTIONS:
Drug: NT-501 ECT implant — NT-501 ECT implant will be placed into the vitreous and out of the visual axis of the study eye. The surgical procedure involves making a small incision through the sclera (white part of the eye), inserting the implant and securing it with a suture.
  Arms: NT-501 ECT Implant
Other: Sham — Sham surgery
  Arms: Sham

SUMMARY:
This is a randomized, sham controlled, masked clinical trial of 60 study participants with glaucoma. Participants with a qualifying study eye will be randomized after screening and baseline evaluations to receive the NT-501 encapsulated cell therapy (ECT) implant or a sham surgery (control arm), and no explant will be required.

An examination for safety will occur one day and one week following implant and periodically thereafter for 24 months post-implant. Based on the primary analysis of data at 6 months, patients in the control arm may be offered the NT-501 ECT implant at the 12 month time point.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet all of the following criteria to join the study (all eligibility criteria must be met at the screening and baseline visits unless otherwise noted):

1. Participant must be medically able to undergo the testing required in the schedule of events (SOE).
2. Participant's clinical diagnosis must be consistent with glaucoma 1. characterized by the following features:

   a) Clinical evidence of progressive retinal ganglion cell (RGC) dysfunction and degeneration using both visual field and at least one structural modality as established by: i. Glaucomatous visual field abnormality. ii. Mean deviation (MD) of -3 to -15 dB. iii. Minimum average retinal nerve fiber layer (RNFL) thickness of 60 μm and maximum average RNFL of 90 μm.

   b) Residual visual field preservation including best-corrected visual acuity (BCVA) better than 20/200 in both eyes.

   c) Two visual field tests of adequate quality with a maximum visual field index (VFI) variability of ± 10%.
3. Participant's glaucoma must be clinically stable, with intraocular pressure (IOP) < 21.
4. If a participant has two eyes meeting study criteria, only the worse eye as determined by visual field index (VFI) will be deemed includable. If both eyes qualify and have the same VFI, a randomization procedure will assign one eye to the study.
5. Participant must understand and sign the informed consent. If the participant's vision is impaired to the point where he/she cannot read the informed consent document, the document will be read to the participant in its entirety.
6. Females of childbearing potential must agree to use an effective form of birth control.
7. Participant must be determined by the presurgical anesthesia or medical team to be fit for ophthalmic surgery for the NT-501 ECT implant insertion.

Exclusion Criteria:

1. Participant is unable to comply with study procedures or follow-up visits.
2. Participant has other optic nerve or retinal degenerative disease causing vision loss, irrespective of whether it is currently treated or untreated.
3. Participant has visual loss to less than 20/200 in non-study eye.
4. Participant is likely to be offered glaucoma surgery within 6 months of screening.
5. Participant has optic nerve atrophy beyond modest pallor.
6. Participant has cataract-associated vision loss to less than 20/40.
7. Participant has a history of ocular herpes zoster.
8. Participant has a requirement of acyclovir and/or related products during study duration. To be eligible for this study, the participant must discontinue use of these products prior to enrollment and must not continue with the products until after they have completed the study.
9. Participant has evidence of corneal opacification or lack of optical clarity.
10. Participant has uveitis or other ocular inflammatory disease.
11. Participant is receiving systemic steroids or other immunosuppressive medications.
12. Participant has diabetic macular edema and/or diabetic retinopathy.
13. Participant has myopic degeneration.
14. Participant is currently participating in or has within the last 3 months participated in any other clinical trial of a drug by ocular or systemic administration.
15. Participant is pregnant or lactating.
16. Participant is on chemotherapy.
17. Participant has a history of malignancy other than basal cell carcinoma, unless it was treated successfully 2 years prior to inclusion in the trial.
18. Participant has, in the opinion of the investigator, any physical or mental condition that would increase the risk of participation in the study or may interfere with the study procedures, evaluations and outcome assessments.
19. Participant has choroidal neovascularization secondary to age related macular degeneration or any other type of retinal degeneration that may interfere with the study procedures, evaluations and outcome assessments.
20. Any intraocular surgery of the study eye within 12 weeks prior to the screening visit
21. History of use of drugs with known retinal toxicity, at retinotoxic doses.
22. Participant has a history or current non-arteritic anterior ischemic neuropathy (NAION)
23. Patient has a history of multiple sclerosis.
24. Participant has glaucoma that is not considered open angle glaucoma, pseudoexfoliation glaucoma or pigmentary glaucoma..

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-06; Primary Completion 2025-08-15 (Actual); Study Completion 2026-08-15 (Estimated)

PRIMARY OUTCOMES:
Visual Field | 6 months
  Determine the efficacy of NT-501 ECT implant in patients with glaucoma as measured by change in visual field through 6 months as assessed by any one of the following three indices:
  1. Visual Field Index (VFI)
  2. Mean Deviation (MD)
  3. Pointwise linear regression (PLR)

SECONDARY OUTCOMES:
Structural measure of retinal ganglion cell layer thickness | 6, 12 and 24 months
  The change in ganglion cell layer thickness as measured by spectral domain optical coherence tomography (sdOCT).
Structural measure of retinal nerve fiber layer thickness | 6, 12 and 24 months
  The change in retinal nerve fiber layer thickness as measured by spectral domain optical coherence tomography (sdOCT).
Contrast sensitivity | 6, 12 and 24 months
  The change in contrast sensitivity through 6, 12 and 24 months
Best corrected visual acuity | 6, 12 and 24 months
  The change in best corrected visual acuity (BCVA) through 6, 12 and 24 months
Optic nerve head structural change | 6, 12 and 24 months
  The change in optic nerve topography as measured by stereo photography through 6, 12, or 24 months 6. The change in visual field as measured by pattern standard deviation (PSD) through 6 months 7. The change in any of the above functional or structural measures at 12 or 24 months
Visual field pattern standard deviation | 6, 12 and 24 months
  The change in visual field as measured by pattern standard deviation (PSD) through 6, 12 or 24 months 7. The change in any of the above functional or structural measures at 12 or 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Byers Eye Institute at Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No